CLINICAL TRIAL: NCT07365670
Title: Comparison of the Best Method for Measuring Anti-Xa Activity in Children Receiving Unfractionated Heparin in Cardiac Intensive Care (COMPAXE-HNF)
Acronym: COMPAXE-HNF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025/RUN/0031; Ethics Committee (Other: CPP Sud Méditerranée I)
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease; Unfractionated Heparin; Anti Xa Activity
Keywords: Unfractionated Heparin; Anti-Xa activity; Pediatric Intensive Care; Congenital Heart Disease; Blood Sampling; Central Venous Catheter; Arterial Catheter; Thrombosis; Hemostasis.
MeSH Terms: conditions — Heart Defects, Congenital; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is an interventional, prospective, single-center (pediatric congenital cardiac intensive care unit at the Réunion University Hospital, North site) study of diagnostic performance.
  * Comparison procedure: sampling from a non-heparinized arterial catheter (gold standard), performed as part of routine care: Method ①
  * Experimental procedure, performed as part of the research: two samples taken from a central venous catheter (CVC)
    * Sample taken from central venous catheter without HNF pause: Method ②
    * Sample taken from central venous catheter with HNF pause: Method ③
  At each anti-Xa activity check in the patients included, the IDE will take the 3 blood samples.
  The order in which samples ② and ③ are taken will be determined by randomization.
  The laboratory will be blinded to the sampling method in order to guarantee the objectivity of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-Xa activity monitoring (Experimental): All patients included in the study
  Interventions: Procedure: blood sampling for measuring anti-Xa activity; Procedure: measurement of anti-XA activity

INTERVENTIONS:
Procedure: blood sampling for measuring anti-Xa activity — Each patient included in the study will have a series of three samples taken every 4 hours for 3 days:
  * Sample taken from a non-heparinized arterial catheter (Gold Standard), performed as part of routine care: Method ①
  * Sample taken from a central venous catheter without stopping the HNF: Method ②
  * Sampling from a central venous catheter with an HNF pause: Method ③
  At each anti-Xa activity check in the included patients, the nurse will take the 3 blood samples.
  The order in which samples ② and ③ are taken will be determined by randomization.
Procedure: measurement of anti-XA activity — Each patient will have, each time that anti-Xa activity needs to be measured, three successive samples taken:
  * Sample taken from a non-heparinized arterial catheter (gold standard), performed as part of routine care: Method ①
  * Sample taken from a central venous catheter without stopping the HNF: Method ②
  * Sample from central venous catheter with HNF pause: Method ③

SUMMARY:
This study aims to compare the accuracy of two different blood sampling methods from a central venous catheter (CVC) for measuring anti-Xa activity in children receiving unfractionated heparin (UFH) from this CVC. The results will be compared to a "gold standard" sample taken from an arterial catheter (KTA) whithout UFH. The objective is to identify a more reliable method for monitoring UFH, thereby reducing the risk of bleeding or thrombosis in these patients.

DETAILED DESCRIPTION:
* Scientific Justification: UFH is widely used in pediatric cardiac intensive care for its short half-life and availability of an antidote. However, monitoring its effect via anti-Xa activity is challenging. The standard method of sampling from a CVC is known to be prone to heparin contamination, leading to inaccurate results (over- or under-anticoagulation). This lack of precision can lead to dangerous complications like major bleeding or thrombotic events. As studies by Palermo et al. (1980) and Bauman et al. (2012) have shown, the unreliability of CVC samples justifies the search for a safer alternative. The arterial catheter (KTA) provides a contamination-free "gold standard," making it the ideal comparison for evaluating the more reliable sampling method.
* Procedure: The study will compare two CVC sampling methods (a standard flush protocol and a new experimental method) against the gold standard (KTA sampling without UFH)
* Follow-up: The study will be conducted over three consecutive days. Each day, three sets of blood samples will be collected every 6 hours per patient (KTA, standard CVC, and experimental CVC).

ELIGIBILITY:
Inclusion Criteria:

* Minors aged 0 to 17 inclusive
* Weight greater than or equal to 3.5 kg
* Admitted to resuscitation or congenital cardiac intensive care
* Requiring treatment with unfractionated heparin at curative doses administered via central venous access
* Equipped with a central arterial and venous catheter
* Affiliated with or beneficiary of a social security scheme
* Free, informed, and written consent signed by one of the two representatives of parental authority and the investigator (no later than the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Newborns < 37 weeks gestation
* Patients treated by a humanitarian organization

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-04-05 (Estimated); Study Completion 2029-04-05 (Estimated)

PRIMARY OUTCOMES:
Measurement of anti-Xa activity (in IU/mL) from two samples (with and without HNF pause) taken from the central venous line where HNF is administered, compared to a sample taken from a non-heparinized arterial catheter (i.e., gold standard). | "From enrollment to the end of study at 72hours"
  Anti-Xa activity and APTT measurements will be performed at the university hospital's central laboratory, which guarantees the consistency of the reagents, automated systems, and techniques used.
  The recommended therapeutic target is between 0.3 and 0.6 IU/mL.

SECONDARY OUTCOMES:
Measurement of APTT from two samples (with and without HNF pause) taken from the central venous line where HNF is administered, compared to a sample taken from a non-heparinized arterial catheter (i.e., gold standard). | "From enrollment to the end of study at 72 hours"
  Activated partial thromboplastin time (APTT):
  Mainly used in the United States and in some French intensive care units, the APTT provides an overall assessment of the activity of several coagulation factors: factor I (or fibrinogen), factor II (or prothrombin), factor V, factor VIII, factor IX, factor X, factor XI, and factor XII. (Figure 1) The APTT is a measure of blood clotting time. It is expressed as a ratio between the patient's APTT and a "control" APTT, which is that of the laboratory. It is expressed in seconds.
  Normal values for the patient APTT/control APTT ratio are between 0.80 s and 1.20 s.
  * Above this range: the risk of bleeding increases.
  * Below this range: treatment is ineffective, with a risk of clot formation.
Measurement of APTT and anti-Xa activity (in IU/mL) from a sample taken from a non-heparinized arterial catheter (i.e., gold standard) | From enrollment to the end of study at 72 hours
  The TCA measurement is performed in the same way.

IPD SHARING:
Plan to Share IPD: No